CLINICAL TRIAL: NCT02400710
Title: Clinician-Supported PTSD Coach vs. Self-Managed PTSD Coach: A Pilot Feasibility Trial
Brief Title: Clinician-Supported PTSD Coach vs. Self-Managed PTSD Coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kyle Possemato, Clinical Research Psychologist, Syracuse VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00615
Record Dates: First submitted 2015-03-16; First posted 2015-03-27 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinician-Supported PTSD Coach (Experimental): Four 20-minute sessions (2 in-person, 2 by phone) focused on instructions for use, setting symptom reductions goals, and assigning specific PTSD Coach activities (i.e., assessments, management strategies, psycho-educational readings) for the participant to complete on their own.
  Interventions: Behavioral: Clinician-Supported PTSD Coach
- Self-Managed PTSD Coach (Active Comparator): One in-person 10-minute session that provides instructions on how to use the PTSD Coach app.
  Interventions: Behavioral: Self-Managed PTSD Coach

INTERVENTIONS:
Behavioral: Clinician-Supported PTSD Coach — Brief primary care-based intervention provided by a mental health clinician who is located in primary care.
  Arms: Clinician-Supported PTSD Coach
Behavioral: Self-Managed PTSD Coach — One 10 minute session explaining how to use the PTSD Coach mobile app.
  Arms: Self-Managed PTSD Coach

SUMMARY:
PTSD Coach is a mobile application (app) that aims to teach individuals self-management strategies for symptoms of Post-traumatic Stress Disorder (PTSD). Despite PTSD Coach's use of evidence-based cognitive behavioral strategies there is still a need to test the effectiveness of the app in managing PTSD symptoms. There is research evidence that self-management programs are often underutilized, but that clinician contact can increase patient involvement. The addition of clinician support may enhance the utilization and effectiveness of the PTSD Coach. In Phase 1 the investigators propose to conduct stakeholder interviews with primary care (PC) and mental health (MH) leadership staff to investigate barriers and facilitators to implementing Clinician-Supported (CS-PTSD Coach) to increase the uptake, use, and impact of PTSD Coach by PC patients. The interviews will inform the development of a CS-PTSD Coach protocol and manual that will be used in phase 2. In phase 2 the investigators propose to conduct a feasibility study where 30 (20 eligible) PC Veterans with diagnostic-level or subthreshold PTSD symptoms will be randomized to receive Self-Managed (SM) PTSD Coach or CS-PTSD Coach. The investigators' specific aims are to 1) investigate the feasibility of recruiting and retaining participants and delivering the SM and CS conditions and 2) conduct a preliminary investigation of the efficacy of SM vs. CS. The investigators predict that CS will lead to greater treatment gains than SM. Effect sizes will be generated for the following outcomes: a) reductions in PTSD, depression, and general distress, and increases in health-related functioning, b) increases in knowledge about PTSD symptoms, PTSD management strategies, and patient coping self-efficacy, c) increases in initiation of tradition PTSD treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in primary care at the Syracuse VAMC,
2. Significant PTSD symptoms. Total PTSD Checklist Score ≥ 40.

Exclusion Criteria:

1. Gross cognitive impairment (as measured by the Blessed Orientation-Memory-Concentration; BOMC)
2. Suicide attempt or intent to commit suicide in the last two months (as measured by the Columbia- Suicide Severity Rating Scale
3. Psychotherapy or mental health counseling for PTSD in the last two months that was received outside of VA primary care
4. A new psychotropic medication or a change in dose of a psychotropic medication for PTSD in the last two months that was received outside of VA primary care
5. Intent to begin PTSD treatment in specialty care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, Ph.D., Principal Investigator — Syracuse VAMC
Locations (1):
- Syracuse VMAC, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinician-Supported PTSD Coach | Self-Managed PTSD Coach
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants completed self-report measures at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician-Supported PTSD Coach | Self-Managed PTSD Coach | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (7.8) | 42.8 (15.4) | 41.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
PTSD Checklist-Specific [Mean (Standard Deviation); unit: units on a scale] — Measures the 17 symptoms of PTSD according to the DSM-IV criteria. Each symptom is measured on a 5-point scale ranging from 1-5, with higher numbers equating to more severe symptoms. Measures range is 17-85. The mean provided is for the total score of all symptoms added together.
  units on a scale | 51.0 (7.7) | 56.0 (15.3) | 53.5 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist-Specific
Description: Measures the 17 symptoms of PTSD according to the DSM-IV. Each symptoms is measured on a 1-5 scale, with higher numbers indicated greater severity. The total range of the scale is 17-85.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinician-Supported PTSD Coach | Self-Managed PTSD Coach
Number analyzed (Participants) | 10 | 10
units on a scale | 40.0 (10.9) | 49.8 (18.1)
Statistical Analysis 1: Comparison: Clinician-Supported PTSD Coach vs Self-Managed PTSD Coach; Test type: Superiority or Other; p = .05, ANOVA

2. Secondary Outcome: Engagement in PTSD Specialty Care as Measured by the Electronic Medical Record
Description: Attendance of at least one session in the PTSD specialty clinic following the completion of the study intervention.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Clinician-Supported PTSD Coach | Self-Managed PTSD Coach
Number analyzed (Participants) | 10 | 10
participants | 7 | 1
Statistical Analysis 1: Comparison: Clinician-Supported PTSD Coach vs Self-Managed PTSD Coach; Test type: Superiority or Other; p = .05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Clinician-Supported PTSD Coach | Self-Managed PTSD Coach
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes